CLINICAL TRIAL: NCT07136844
Title: Gait Analysis Parameter and Upper Limb Evaluation in Adult Patients With Neurological or Metabolic Pathology
Acronym: Acti-Adult
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other); SYSNAV (Industry)
Responsible Party: Principal Investigator, Laurent Servais, Principal Investigator, Pediatrician, Centre Hospitalier Universitaire de Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ActiLiège Adult
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Neuromuscular Diseases; Obesity (Disorder); Myotonic Dystrophy 1; Myasthenic Syndrome; Charcot Marie Tooth Disease (CMT); Glycogen Storage Disease Type II Pompe Disease; Facio-Scapulo-Humeral Dystrophy; Myasthenia Gravis; Huntington Disease; Progressive Supranuclear Palsy (PSP); Hereditary Spastic Paraplegia; Ataxia, Spinocerebellar
MeSH Terms: conditions — Neuromuscular Diseases; Obesity; Myotonic Dystrophy; Lambert-Eaton Myasthenic Syndrome; Charcot-Marie-Tooth Disease; Muscular Dystrophy, Facioscapulohumeral; Myasthenia Gravis; Huntington Disease; Supranuclear Palsy, Progressive; Spastic Paraplegia, Hereditary; Spinocerebellar Ataxias | interventions — Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Neuromuscular condition - Muscle disease (Experimental)
  Interventions: Device: Syde; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Other: Patient's Global Impression of Change (PGIC)
- Neuromuscular condition - Neuropathy (Experimental)
  Interventions: Device: Syde; Diagnostic Test: Dynamometric measurements of muscle strength; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Diagnostic Test: The Charcot-Marie-Tooth examination score (CMTES); Diagnostic Test: 9-Hole Peg Test (9-HPT); Other: Patient's Global Impression of Change (PGIC)
- Ataxia (Experimental)
  Interventions: Device: Syde; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Diagnostic Test: 9-Hole Peg Test (9-HPT); Diagnostic Test: The Scale for the Assessment and Rating of Ataxia (SARA); Other: Patient's Global Impression of Change (PGIC)
- Huntington disease (HD) and HD-like (Experimental)
  Interventions: Device: Syde; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Diagnostic Test: The Unified Huntington's Disease Rating Scale (UHDRS); Other: Patient's Global Impression of Change (PGIC)
- Progressive supranuclear palsy (PSP) and PSP-like (Experimental)
  Interventions: Device: Syde; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Diagnostic Test: The Timed up and go test (TUG); Diagnostic Test: The Progressive Supranuclear Palsy Rating Scale (PSP-RS); Diagnostic Test: The Montreal Cognitive Assessment (MOCA); Other: Patient's Global Impression of Change (PGIC)
- Spastic paraplesia and conditions where spasticity predominates, incl. stroke (Experimental)
  Interventions: Device: Syde; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Other: Patient's Global Impression of Change (PGIC)
- Obese patients (Experimental)
  Interventions: Device: Syde; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Other: Patient's Global Impression of Change (PGIC)
- Neuromuscular condition - Neuromuscular Junction (Experimental)
  Interventions: Device: Syde; Diagnostic Test: The 6-minute walk test (6MWT); Diagnostic Test: The 10-meter test (10MWT); Diagnostic Test: The 4 stair-climbing test (4SC); Diagnostic Test: Test of rising from the floor (TRF); Diagnostic Test: Quantitative Myasthenia Gravis (QMG); Diagnostic Test: The Myasthenia Gravis Activities of Daily Living Scale (MG-ADL); Other: Patient's Global Impression of Change (PGIC)

INTERVENTIONS:
Device: Syde — Syde is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.
Diagnostic Test: Dynamometric measurements of muscle strength — Dynamometric measurements of the maximum force of the following functions will be taken with the MyoTools: palmar grip (MyoGrip) and thumb-index pinch (MyoPinch). Test will be realized on the dominant side. Patients will be encouraged during the test. They will be given three trials and the best score will be entered.
  Arms: Neuromuscular condition - Neuropathy
Diagnostic Test: The 6-minute walk test (6MWT) — This test consists of covering the greatest possible distance within 6 minutes, walking back and forth along a 25-meter hallway. The subject may stop if they need to. The evaluator will record the elapsed time after each half-lap, and the final distance that was covered at the end of the test. No help will be allowed during the test.
Diagnostic Test: The 10-meter test (10MWT) — During this test, the subject must cover a distance of 10 meters as rapidly as possible. This test will be performed 3 times. The participant will be allowed to rest for one minute after the first and second instances of the test. No help will be allowed during the test.
Diagnostic Test: The 4 stair-climbing test (4SC) — This is a standardized test during which the subject must climb the 4 stair steps as rapidly as possible. This test will be performed 3 times. The participant will be allowed to rest for one minute after the first and second instances of the test, or more if needed.
Diagnostic Test: Test of rising from the floor (TRF) — This is a standardized test during which the subject must rise from the floor as rapidly as possible. The test starts with the participant lying on their back. This test will be performed 3 times. The participant will be allowed to rest for one minute after the first and second instances of the test.
Diagnostic Test: The Timed up and go test (TUG) — During this standardized test, the subject is observed and timed while he/she rises from a chair, walks 3 meters, performs a 180° turn, walk back toward the chair and sits down.
  Arms: Progressive supranuclear palsy (PSP) and PSP-like
Diagnostic Test: The Progressive Supranuclear Palsy Rating Scale (PSP-RS) — This 28-item clinician-rated scale assesses motor and non-motor symptom severity in patients with PSP, with a score ranging from 0 (normal) to 100.
  Arms: Progressive supranuclear palsy (PSP) and PSP-like
Diagnostic Test: The Montreal Cognitive Assessment (MOCA) — The MOCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive function, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Scores on the MOCA range from 0 to 30, with higher score being better outcome.
  Arms: Progressive supranuclear palsy (PSP) and PSP-like
Diagnostic Test: The Charcot-Marie-Tooth examination score (CMTES) — The CMTES is a 28-point composite score that rates the patient's symptoms and signs. It is part of the Charcot-Marie-Tooth (CMT) neuropathy score and has been validated as a reproducible measure of disability in CMT. Higher scores indicate more severe neuropathy.
  Arms: Neuromuscular condition - Neuropathy
Diagnostic Test: 9-Hole Peg Test (9-HPT) — The 9-HPT is a quantitative test of upper limb function. It is the second component of the Multiple Sclerosis Functional Composite (MSFC). The patient sits at a table with a shallow container containing nine sticks and a wooden or plastic block containing nine empty holes. When a timer is started, the patient places the nine sticks one after the other as quickly as possible into the nine holes and, once they are all in the holes, removes them as quickly as possible. The total time taken to complete the task is recorded. Two consecutive attempts with the dominant hand are immediately followed by two consecutive attempts with the non-dominant hand.
  Arms: Ataxia; Neuromuscular condition - Neuropathy
Diagnostic Test: The Unified Huntington's Disease Rating Scale (UHDRS) — This 74-item clinical rating scale assesses patient performance and capacity in 4 domains: motor function, cognitive function, behavioral abnormalities, and functional capacity.
  Arms: Huntington disease (HD) and HD-like
Diagnostic Test: Quantitative Myasthenia Gravis (QMG) — The QMG is a clinician-rated 13-item scale used to quantify disease severity in patients with MG. The scale grades each domain (ocular, bulbar, respiratory, and limb function), with a total score ranging from 0 to 39 (lower score indicating a better clinical outcome).
  Arms: Neuromuscular condition - Neuromuscular Junction
Diagnostic Test: The Myasthenia Gravis Activities of Daily Living Scale (MG-ADL) — This is an 8-item patient-reported scale assessing MG symptoms and their effects on daily activities. The score ranges from 0 to 24, with higher score indicating a worse clinical outcome.
  Arms: Neuromuscular condition - Neuromuscular Junction
Diagnostic Test: The Scale for the Assessment and Rating of Ataxia (SARA) — This 8-item scale was developed to assess ataxia severity and disease progression. It evaluates gait and balance, speech, and upper and lower limb coordination. The score ranges from 0 to 40, with higher score indicating a worse clinical outcome.
  Arms: Ataxia
Other: Patient's Global Impression of Change (PGIC) — PGIC is a patient-reported scale used to assess how a patient feels their condition has changed over time. It typically uses a 7-point scale to capture the patient's overall perception of improvement in symptoms, function, and quality of life.

SUMMARY:
The ActiLiège-Adult study is a prospective, longitudinal, observational study designed to collect natural history data on adult patients with neurological or metabolic diseases affecting movement. Conducted at the Centre de Référence Liégeois des Maladies Neuromusculaires in Liège, Belgium, the study will enroll 300 ambulant patients, including individuals with neuromuscular disorders and obesity. Using the Syde® wearable device, the study aims to continuously monitor motor function in real-life settings over a period of up to two years. The primary objective is to evaluate the utility of digital mobility outcomes, such as the 95th centile of stride velocity (SV95C), as reliable and objective endpoints for future clinical trials.

DETAILED DESCRIPTION:
Following the qualification of the 95th centile of stride velocity (SV95C) as a primary digital endpoint in Duchenne muscular dystrophy (DMD), there is growing interest in extending such digital assessments to other neurological and metabolic diseases that impair movement. Traditional in-clinic functional tests (e.g., 6-minute walk test, 10-meter walk/run) provide only limited snapshots of motor ability and are influenced by external factors such as motivation and fatigue. Similarly, motor function scales and biomarkers, while useful, often lack objectivity or established clinical relevance.

The ActiLiège-Adult study aims to address these limitations by leveraging the Syde® device, a wearable magneto-inertial sensor worn on the wrist and/or ankle, to continuously monitor motor activity in daily life. This device has been previously validated in DMD and other neuromuscular conditions and has been used in both interventional and natural history studies.

This academic study will enroll 300 ambulant adult patients, including 220 with neurological diseases and 20 with obesity, with a minimum of 20 patients per disease type. Ambulation is defined as the ability to walk 10 meters unaided. Patients who lose ambulation during the study will continue to be followed with adapted assessments.

Participants will be monitored for up to two years (six months for diseases affecting the neuromuscular junction). Standardized clinical assessments-including timed tests, motor function evaluations, and strength measurements-will be conducted at baseline and every six months. These will be compared with continuous data collected by the Syde® device. Additionally, patients will complete a Patient Global Impression of Change (PGI-C) questionnaire every six months.

The study's goal is to generate robust, real-world data to support the development of objective, sensitive, and clinically meaningful digital endpoints for use in future therapeutic trials targeting movement disorders.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant patients (i.e. able to walk 10 meters without assistance)
* Confirmed diagnosis by the investigator based on current gold standard in his/her disease (genetic testing, clinical criteria, etc.)

  * Myotonic dystrophy type 1 (DM1) and Charcot-Marie-Tooth (CMT) patients should present sensitive of motor signs on physical examination.
  * Myasthenic patients should be seropositive, and Myasthenia Gravis Foundation of America (MGFA) class II to IV.
  * Patient with morbid obesity (Body Mass Index> or = 35 at inclusion visit).
* Signed informed consent form by patient him/herself and patient willing and able to comply with all study procedures.

Exclusion Criteria:

* Non-ambulant patients
* Patients with extreme cognitive disorders that limit their understanding of the exercises to be performed
* Patients who have undergone a surgical procedure or who have experienced recent trauma (within fewer than 6 months) affecting the upper or lower limbs
* A concomitant chronic or acute neurological, endocrine, infectious, allergic, or inflammatory pathology within the 3-week period immediately prior to inclusion
* Patients who are participating in an interventional clinical trial
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
95th Centile of Stride Velocity (SV95C) | Every 6 months for up to 2 years
  Change in SV95C as measured by the Syde® wearable device, used to assess ambulatory function in real-life settings.

SECONDARY OUTCOMES:
Device Acceptability and Adherence | Over 2 years
  Measures of user engagement with the Syde® device over time, including total recording time, valid days (≥5 hours), and time to reach 50 and 180 hours.
Correlation between Syde® and 6MWT | Every 6 months for up to 2 years
  Correlation between the Syde digital variable and results from the 6-minute walk test (6MWT)
Correlation between Syde® and 10MWT | Every 6 months for up to 2 years
  Correlation between the Syde digital variable and results from the 10-meter test (10MWT)
Correlation between Syde® and 4SC | Every 6 months for up to 2 years
  Correlation between the Syde digital variable and results from the 4 stair-climbing test (4SC)
Correlation between Syde® and TRF | Every 6 months for up to 2 years
  Correlation between the Syde digital variable and results from the test of rising from the floor (TRF)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- Centre de référence des maladies neuromusculaire, Centre Hospitalier Régional de la Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No